CLINICAL TRIAL: NCT02268214
Title: A Multicenter, Randomized, Double-Blind, Placebo-controlled, Parallel Group, Phase 3 Study to Evaluate the Efficacy and Safety of Dapagliflozin as an Add-on to Insulin Therapy in Subjects With Type 1 Diabetes Mellitus
Brief Title: Dapagliflozin Evaluation in Patients With Inadequately Controlled Type 1 Diabetes
Acronym: DEPICT 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MB102-229; 2013-004674-97 (EudraCT Number); D1695C00006 (Other: AstraZenenca)
Record Dates: First submitted 2014-10-15; First posted 2014-10-20 (Estimated); Results first posted 2018-03-29 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-08

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Dapagliflozin; Efficacy; Safety; Add on to insulin; Oral Antidiabetic; Type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A: Dapagliflozin (Experimental): Dapagliflozin 5 mg tablet orally, once daily for 52 weeks
  Interventions: Drug: Dapagliflozin
- Arm B: Dapagliflozin (Experimental): Dapagliflozin 10 mg tablet orally, once daily for 52 weeks
  Interventions: Drug: Dapagliflozin
- Arm C: Placebo for Dapagliflozin (Placebo Comparator): Placebo tablet orally, once daily for 52 weeks
  Interventions: Drug: Placebo for dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin — Tablets
  Arms: Arm A: Dapagliflozin; Arm B: Dapagliflozin
Drug: Placebo for dapagliflozin — Tablets
  Arms: Arm C: Placebo for Dapagliflozin

SUMMARY:
The purpose of this study is to determine if adding dapagliflozin to insulin is a safe and effective therapy to improve glycemic control in patients with type 1 diabetes.

DETAILED DESCRIPTION:
Study Classification: Safety, Efficacy and Pharmacokinetics/dynamics

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 1 Diabetes mellitus (T1DM)
* Central laboratory C-peptide < 0.7 ng/ml (0.23 nmol/L)
* Insulin use for at least 12 months per patient reported or medical records
* Method of insulin administration (MDI or CSII) must have been unchanged for at least 3 months prior to screening
* Subjects must be on a total insulin dose of ≥ 0.3 U/kg/day for at least 3 months prior to screening
* If on MDI insulin administration, subject must be on ≥ 3x injections per day
* Screening Visit: Central laboratory HbA1c ≥ 7.7% and ≤ 11.0%
* Body mass index (BMI) ≥ 18.5 kg/m2

Exclusion Criteria:

* History of Type 2 Diabetes mellitus (T2DM) or maturity onset diabetes of the young (MODY), pancreatic surgery, or chronic pancreatitis that could result in decreased beta cell capacity
* Taking metformin and/or thiazolidinediones within 2 months prior to screening
* Taking any antidiabetic medication (other than insulin), within 1 month prior to screening

  - Taking GLP-1 receptor agonist within 2 months prior to screening for once weekly administration and within 1 month prior to screening for once or twice daily administration
* History of diabetes ketoacidosis requiring medical intervention within 1 month prior to screening
* History of hospital admission for glycemic control (either hyperglycemia or hypoglycemia) within 1 month prior to screening
* Frequent episodes of severe hypoglycemia (more than one episode requiring medical assistance, emergency care), and/or glucagon therapy administered by a third-party individual within 1 month prior to screening
* History of Addison's disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 833 (Actual)
Dates: Start 2014-11-11 (Actual); Primary Completion 2017-01-04 (Actual); Study Completion 2017-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Maria Langkilde, Study Director — AstraZeneca
Locations (127):
- United States (36):
  - Research Site, Little Rock, Arkansas
  - Research Site, Encino, California
  - Research Site, La Mesa, California
  - Research Site, San Diego, California
  - Research Site, Tarzana, California
  - Research Site, Torrance, California
  - Research Site, Aurora, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Cooper City, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Port Orange, Florida
  - Research Site, Idaho Falls, Idaho
  - Research Site, Des Moines, Iowa
  - Research Site, Louisville, Kentucky
  - Research Site, Portland, Maine
  - Research Site, Hyattsville, Maryland
  - Research Site, Rockville, Maryland
  - Research Site, Kalamazoo, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Chesterfield, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Albany, New York
  - Research Site, Buffalo, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Greenville, North Carolina
  - Research Site, Morehead City, North Carolina
  - Research Site, Langhorne, Pennsylvania
  - Research Site, Kingsport, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Amarillo, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Olympia, Washington
- Australia (7):
  - Research Site, Concord
  - Research Site, Daw Park
  - Research Site, Fitzroy
  - Research Site, Heidelberg West
  - Research Site, Newcastle
  - Research Site, Southport
  - Research Site, Wollongong
- Austria (3):
  - Research Site, Innsbruck
  - Research Site, Saint Stefan/Stainz
  - Research Site, Vienna
- Belgium (3):
  - Research Site, Bonheiden
  - Research Site, Leuven
  - Research Site, Liège
- Canada (4):
  - Research Site, Vancouver, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, London, Ontario
  - Research Site, Laval, Quebec
- Denmark (4):
  - Research Site, Arhus C
  - Research Site, Esbjerg
  - Research Site, Odense
  - Research Site, Randers NØ
- Finland (5):
  - Research Site, Helsinki
  - Research Site, Jyväskylä
  - Research Site, Kuopio
  - Research Site, Oulu
  - Research Site, Tampere
- France (5):
  - Research Site, Besançon
  - Research Site, Corbeil-Essonnes
  - Research Site, Dijon
  - Research Site, Saint-Herblain
  - Research Site, Vandœuvre-lès-Nancy
- Germany (12):
  - Research Site, Aschaffenburg
  - Research Site, Aßlar
  - Research Site, Bad Oeynhausen
  - Research Site, Falkensee
  - Research Site, Munich
  - Research Site, Münster
  - Research Site, Neuwied
  - Research Site, Oldenburg
  - Research Site, Pohlheim
  - Research Site, Schweinfurt
  - Research Site, Sulzbach
  - Research Site, Witten
- Hungary (6):
  - Research Site, Baja
  - Research Site, Balatonfüred
  - Research Site, Budapest
  - Research Site, Létavértes
  - Research Site, Szeged
  - Research Site, Zalaegerszeg
- Israel (5):
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Safed
  - Research Site, Tel Aviv
  - Research Site, Tikva
- Italy (7):
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Padowa
  - Research Site, Palermo
  - Research Site, Ravenna
  - Research Site, Sesto San Giovanni
  - Research Site, Siena
- Mexico (10):
  - Research Site, Aguascalientes
  - Research Site, Chihuahua City
  - Research Site, Cuernavaca
  - Research Site, Guadalajara
  - Research Site, Mérida
  - Research Site, México
  - Research Site, Monterrey
  - Research Site, Torreón
  - Research Site, Zapopan
  - Research Site, Zapopan, Jalisco
- Romania (5):
  - Research Site, Bucharest
  - Research Site, Dolj
  - Research Site, Galati
  - Research Site, Iași
  - Research Site, Timișoara
- Spain (5):
  - Research Site, A Coruña
  - Research Site, Almería
  - Research Site, Barcelona
  - Research Site, Seville
  - Research Site, Valencia
- Sweden (4):
  - Research Site, Gothenburg
  - Research Site, Karlstad
  - Research Site, Lund
  - Research Site, Uppsala
- United Kingdom (6):
  - Research Site, Belfast
  - Research Site, Chesterfield
  - Research Site, Dundee
  - Research Site, Nottingham
  - Research Site, Sheffield
  - Research Site, Welwyn Garden City

REFERENCES:
- [Derived] Nardone M, Kugathasan L, Sridhar VS, Dutta P, Campbell DJT, Layton AT, Perkins BA, Barbour S, Lam TKT, Levin A, Lovblom LE, Mucsi I, Rabasa-Lhoret R, Rac VE, Senior P, Sigal RJ, Stanimirovic A, Persson F, Stougaard EB, Doria A, Cherney DZI. Modeling Cardiorenal Protection with Sodium-Glucose Cotransporter 2 Inhibition in Type 1 Diabetes: An Analysis of DEPICT-1 and DEPICT-2. Clin J Am Soc Nephrol. 2025 Apr 1;20(4):529-538. doi: 10.2215/CJN.0000000641. Epub 2025 Feb 7. PMID 39918875
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Melin J, Tang W, Rekic D, Hamren B, Penland RC, Boulton DW, Parkinson J. Dapagliflozin Pharmacokinetics Is Similar in Adults With Type 1 and Type 2 Diabetes Mellitus. J Clin Pharmacol. 2022 Oct;62(10):1227-1235. doi: 10.1002/jcph.2062. Epub 2022 May 2. PMID 35403243
- [Derived] Groop PH, Dandona P, Phillip M, Gillard P, Edelman S, Jendle J, Xu J, Scheerer MF, Thoren F, Iqbal N, Repetto E, Mathieu C. Effect of dapagliflozin as an adjunct to insulin over 52 weeks in individuals with type 1 diabetes: post-hoc renal analysis of the DEPICT randomised controlled trials. Lancet Diabetes Endocrinol. 2020 Oct;8(10):845-854. doi: 10.1016/S2213-8587(20)30280-1. PMID 32946821
- [Derived] Mathieu C, Dandona P, Birkenfeld AL, Hansen TK, Iqbal N, Xu J, Repetto E, Scheerer MF, Thoren F, Phillip M. Benefit/risk profile of dapagliflozin 5 mg in the DEPICT-1 and -2 trials in individuals with type 1 diabetes and body mass index >/=27 kg/m2. Diabetes Obes Metab. 2020 Nov;22(11):2151-2160. doi: 10.1111/dom.14144. Epub 2020 Aug 20. PMID 32691513
- [Derived] Parkinson J, Tang W, Astrand M, Melin J, Ekholm E, Hamren B, Boulton DW. Model-based characterization of the relationship between dapagliflozin systemic exposure and HbA1c response in patients with type 1 diabetes mellitus. Diabetes Obes Metab. 2019 Jun;21(6):1381-1387. doi: 10.1111/dom.13664. Epub 2019 Mar 14. PMID 30756462
- [Derived] Dandona P, Mathieu C, Phillip M, Hansen L, Tschope D, Thoren F, Xu J, Langkilde AM; DEPICT-1 Investigators. Efficacy and Safety of Dapagliflozin in Patients With Inadequately Controlled Type 1 Diabetes: The DEPICT-1 52-Week Study. Diabetes Care. 2018 Dec;41(12):2552-2559. doi: 10.2337/dc18-1087. Epub 2018 Oct 23. PMID 30352894
- [Derived] Dandona P, Mathieu C, Phillip M, Hansen L, Griffen SC, Tschope D, Thoren F, Xu J, Langkilde AM; DEPICT-1 Investigators. Efficacy and safety of dapagliflozin in patients with inadequately controlled type 1 diabetes (DEPICT-1): 24 week results from a multicentre, double-blind, phase 3, randomised controlled trial. Lancet Diabetes Endocrinol. 2017 Nov;5(11):864-876. doi: 10.1016/S2213-8587(17)30308-X. Epub 2017 Sep 14. PMID 28919061
- See also: MB102229_CSP — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3676&filename=MB102229-revprot2_1_15.08.17_Redacted.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was enrolled on 11 November 2014. The last subject completed the 24-week short-term treatment period 04 January 2017 and the last subject completed the study 25 August 2017. This study was conducted at 138 sites in 17 countries.
Pre-assignment Details: 833 participants were randomized to a treatment group. Of the 771 participants not randomized to a treatment group: 585 No longer met study criteria, 125 withdrew consent, 26 were lost to follow-up, and 35 did not continue for other reasons
Groups:
- Dapagliflozin 5 mg + Insulin: Dapagliflozin 5 mg oral tablet once daily + background insulin
- Dapagliflozin 10 mg + Insulin: Dapagliflozin 10 mg oral tablet once daily + background insulin
- Placebo + Insulin: Placebo oral tablet once daily + background insulin
Period: Overall Study
Arm/Group | Dapagliflozin 5 mg + Insulin | Dapagliflozin 10 mg + Insulin | Placebo + Insulin
Started | 277 | 296 | 260
COMPLETED 24 WEEK PERIOD | 252 | 273 | 232
Completed | 235 | 255 | 218
Not Completed | 42 | 41 | 42
Not completed — Subject no longer meets study criteria | 0 | 2 | 0
Not completed — Pregnancy | 2 | 2 | 1
Not completed — Lost to Follow-up | 3 | 3 | 4
Not completed — Lack of Efficacy | 1 | 0 | 2
Not completed — Adverse Event | 11 | 14 | 9
Not completed — Withdrawal by Subject | 4 | 5 | 10
Not completed — Subject request to discontinue treatment | 10 | 8 | 6
Not completed — Poor/non-compliance | 2 | 1 | 2
Not completed — Other reasons | 7 | 3 | 3
Not completed — Not entering long-term period | 2 | 3 | 5

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: It consists of all subjects who received at least one dose of double-blind study medication during the short-term double-blind treatment period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin 5 mg + Insulin | Dapagliflozin 10 mg + Insulin | Placebo + Insulin | Total
Number analyzed (Participants) | 277 | 296 | 260 | 833
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.1 (13.94) | 43.4 (13.89) | 42.7 (13.57) | 42.7 (13.80)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 262 | 279 | 246 | 787
  Between 65 and 75 years | 15 | 16 | 14 | 45
  >= 75 years | 0 | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 158 | 144 | 128 | 430
  Male | 119 | 152 | 132 | 403

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change in HbA1c From Baseline at Week 24
Description: Adjusted mean change from baseline in HbA1c at Week 24 (Repeated Measures Model[RMM]).
Time Frame: From Baseline to Week 24
Population: All randomized subjects who took at least one dose of double-blind study medication during the short-term double-blind period. The first 55 randomized subjects will be excluded from the full analysis dataset due to the presence of a randomization system error.
Measure: Least Squares Mean (Standard Error); unit: Percentage of hemoglobin
Arm/Group | Dapagliflozin 5 mg + Insulin | Dapagliflozin 10 mg + Insulin | Placebo + Insulin
Number analyzed (Participants) | 254 | 254 | 257
Percentage of hemoglobin | -0.45 (0.0537) | -0.47 (0.0538) | -0.03 (0.0540)
Statistical Analysis 1: Comparison: Dapagliflozin 5 mg + Insulin vs Placebo + Insulin; Test type: Superiority; p < 0.0001, RMM; Repeated Measures Model; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-0.56 to -0.28], Standard Error of Mean 0.0697
Statistical Analysis 2: Comparison: Dapagliflozin 10 mg + Insulin vs Placebo + Insulin; Test type: Superiority; p < 0.0001, RMM; Repeated Measures Model; Median Difference (Final Values) = -0.45, 95% CI 2-sided [-0.58 to -0.31], Standard Error of Mean 0.0696

2. Secondary Outcome: Adjusted Mean Percent Change in Total Daily Insulin Dose From Baseline at Week 24
Description: Adjusted mean change from baseline in Total Daily Insulin Dose at Week 24 (Repeated Measures Model[RMM])
Time Frame: From Baseline to Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: IU
Arm/Group | Dapagliflozin 5 mg + Insulin | Dapagliflozin 10 mg + Insulin | Placebo + Insulin
Number analyzed (Participants) | 258 | 254 | 258
IU | -7.74 (1.4881) | -12.16 (1.4326) | 1.16 (1.6593)
Statistical Analysis 1: Comparison: Dapagliflozin 5 mg + Insulin vs Placebo + Insulin; Test type: Superiority; p < 0.0001, RMM; Repeated Measures Model; Mean Difference (Final Values) = -8.80, 95% CI 2-sided [-12.56 to -4.88], Standard Error of Mean 1.9555
Statistical Analysis 2: Comparison: Dapagliflozin 10 mg + Insulin vs Placebo + Insulin; Test type: Superiority; p < 0.0001, RMM; Repeated Measures Model; Mean Difference (Final Values) = -13.17, 95% CI 2-sided [-16.75 to -9.43], Standard Error of Mean 1.8643

3. Secondary Outcome: Adjusted Mean Percent Change in Body Weight From Baseline at Week 24
Description: Adjusted mean percent change from baseline in body weight at Week 24 (Repeated Measures Model[RMM])
Time Frame: From Baseline to Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Kg
Arm/Group | Dapagliflozin 5 mg + Insulin | Dapagliflozin 10 mg + Insulin | Placebo + Insulin
Number analyzed (Participants) | 259 | 258 | 259
Kg | -3.00 (0.2330) | -3.67 (0.2299) | 0.05 (0.2407)
Statistical Analysis 1: Comparison: Dapagliflozin 5 mg + Insulin vs Placebo + Insulin; Test type: Superiority; p < 0.0001, RMM; Repeated Measures Model; Mean Difference (Final Values) = -3.05, 95% CI 2-sided [-3.68 to -2.41], Standard Error of Mean 0.3251
Statistical Analysis 2: Comparison: Dapagliflozin 10 mg + Insulin vs Placebo + Insulin; Test type: Superiority; p < 0.0001, RMM; Repeated Measures Model; Mean Difference (Final Values) = -3.72, 95% CI 2-sided [-4.34 to -3.08], Standard Error of Mean 0.3213

4. Secondary Outcome: Adjusted Mean Change in 24-hour Mean Continuous Glucose Monitoring Glucose From Baseline at Week 24
Description: Adjusted mean change in 24-hour mean Continuous Glucose Monitoring glucose from baseline at Week 24 (Repeated Measures Model[RMM])
Time Frame: From Baseline to Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Dapagliflozin 5 mg + Insulin | Dapagliflozin 10 mg + Insulin | Placebo + Insulin
Number analyzed (Participants) | 238 | 239 | 234
mg/dL | -10.28 (1.8862) | -12.97 (1.9231) | 5.06 (1.9320)
Statistical Analysis 1: Comparison: Dapagliflozin 5 mg + Insulin vs Placebo + Insulin; Test type: Superiority; p < 0.0001, RMM; Repeated Measures Model; Mean Difference (Final Values) = -15.34, 95% CI 2-sided [-20.22 to -10.46], Standard Error of Mean 2.4859
Statistical Analysis 2: Comparison: Dapagliflozin 10 mg + Insulin vs Placebo + Insulin; Test type: Superiority; p < 0.0001, RMM; Repeated Measures Model; Mean Difference (Final Values) = -18.03, 95% CI 2-sided [-22.95 to -13.11], Standard Error of Mean 2.5050

5. Secondary Outcome: Adjusted Mean Change in 24-hour Continuous Glucose Monitoring MAGE From Baseline at Week 24
Description: Adjusted Mean Change in 24-hour Continuous Glucose Monitoring Mean Amplitude of Glucose Excursions (MAGE) from Baseline at Week 24 (Repeated Measures Model[RMM])
Time Frame: From Baseline to Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Dapagliflozin 5 mg + Insulin | Dapagliflozin 10 mg + Insulin | Placebo + Insulin
Number analyzed (Participants) | 238 | 239 | 234
mg/dL | -14.92 (1.9915) | -16.55 (2.0419) | 2.38 (2.0477)
Statistical Analysis 1: Comparison: Dapagliflozin 5 mg + Insulin vs Placebo + Insulin; Test type: Superiority; p < 0.0001, RMM; Repeated Measures Model; Mean Difference (Final Values) = -17.30, 95% CI 2-sided [-22.46 to -12.14], Standard Error of Mean 2.6273
Statistical Analysis 2: Comparison: Dapagliflozin 10 mg + Insulin vs Placebo + Insulin; Test type: Superiority; p < 0.0001, RMM; Repeated Measures Model; Mean Difference (Final Values) = -18.93, 95% CI 2-sided [-24.13 to -13.73], Standard Error of Mean 2.6482

6. Secondary Outcome: Adjusted Mean Change in Percent 24-hour Continuous Glucose Monitoring Glucose > 70 and <= 180 (mg/dL) From Baseline at Week 24
Description: Adjusted Mean Change in Percent 24-hour Continuous Glucose Monitoring Glucose > 70 and <= 180 (mg/dL) from Baseline at Week 24 (Repeated Measures Model[RMM])
Time Frame: From Baseline to Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | Dapagliflozin 5 mg + Insulin | Dapagliflozin 10 mg + Insulin | Placebo + Insulin
Number analyzed (Participants) | 238 | 239 | 234
Percentage | 6.98 (0.8824) | 8.52 (0.9000) | -2.13 (0.9032)
Statistical Analysis 1: Comparison: Dapagliflozin 5 mg + Insulin vs Placebo + Insulin; Test type: Superiority; p < 0.0001, RMM; Repeated Measures Model; Mean Difference (Final Values) = 9.11, 95% CI 2-sided [6.83 to 11.39], Standard Error of Mean 1.1611
Statistical Analysis 2: Comparison: Dapagliflozin 10 mg + Insulin vs Placebo + Insulin; Test type: Superiority; p < 0.0001, RMM; Repeated Measures Model; Mean Difference (Final Values) = 10.65, 95% CI 2-sided [8.35 to 12.94], Standard Error of Mean 1.1689

7. Secondary Outcome: Subjects With HbA1c Reduction From Baseline to Week 24 (LOCF) >= 0.5% and Without Severe Hypoglycemia Events
Description: Subjects with HbA1c reduction from baseline to week 24 (LOCF) >= 0.5% and without severe hypoglycemia events
Time Frame: From Baseline to Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dapagliflozin 5 mg + Insulin | Dapagliflozin 10 mg + Insulin | Placebo + Insulin
Number analyzed (Participants) | 256 | 254 | 257
Participants
  Responders | 127 | 129 | 65
Statistical Analysis 1: Comparison: Dapagliflozin 5 mg + Insulin vs Placebo + Insulin; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 3.09, 95% CI 2-sided [2.10 to 4.56], Standard Error of Mean 0.1980
Statistical Analysis 2: Comparison: Dapagliflozin 10 mg + Insulin vs Placebo + Insulin; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 3.29, 95% CI 2-sided [2.23 to 4.85], Standard Error of Mean 0.1979

ADVERSE EVENTS:
Time Frame: Onset on or after the first date of double-blind treatment and on or prior to the last day of treatment 24-week short-term period, 28-week extension period and the 30-day folllow-up period
Description: Participants were questioned at each study visit about the occurrence of any health problems and any examination conducted at a study visit was assessed in comparison to the status at study entry.
Arm/Group | Dapagliflozin 5 mg + Insulin | Dapagliflozin 10 mg + Insulin | Placebo + Insulin
All-Cause Mortality (participants affected / at risk) | 0/277 | 0/296 | 1/260
Serious Adverse Events (participants affected / at risk) | 37/277 | 40/296 | 30/260
Other Adverse Events (participants affected / at risk) | 123/277 | 118/296 | 99/260
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin 5 mg + Insulin (N=277) | Dapagliflozin 10 mg + Insulin (N=296) | Placebo + Insulin (N=260)
Myocardial infarction (Cardiac disorders) | 0 | 1 (1) | 0
Angina pectoris (Cardiac disorders) | 1 (1) | 0 | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 | 1 (1) | 0
Blindness unilateral (Eye disorders) | 1 (1) | 0 | 0
Cataract (Eye disorders) | 1 (1) | 0 | 0
Vitreous haemorrhage (Eye disorders) | 2 (3) | 0 | 0
Gastrointestinal hypomotility (Gastrointestinal disorders) | 0 | 1 (1) | 0
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1 (1) | 0
Chest pain (General disorders) | 1 (1) | 2 (2) | 1 (1)
Impaired healing (General disorders) | 0 | 1 (1) | 0
Hyperparathyroidism primary (Endocrine disorders) | 0 | 0 | 1 (1)
Ophthalmoplegia (Eye disorders) | 0 | 0 | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 | 1 (1) | 0
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 | 1 (1) | 0
Pyrexia (General disorders) | 0 | 0 | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 (1) | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 (1) | 0
Cyclic vomiting syndrome (Gastrointestinal disorders) | 0 | 1 (1) | 0
Diabetic gastroparesis (Gastrointestinal disorders) | 1 (2) | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 (1)
Hepatic haematoma (Hepatobiliary disorders) | 1 (1) | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 1 (1)
Bronchitis (Infections and infestations) | 0 | 0 | 1 (1)
Cellulitis (Infections and infestations) | 0 | 0 | 1 (1)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 | 0
Influenza (Infections and infestations) | 0 | 1 (1) | 0
Localised infection (Infections and infestations) | 1 (1) | 0 | 0
Nasal abscess (Infections and infestations) | 0 | 0 | 1 (1)
Perineal abscess (Infections and infestations) | 0 | 0 | 1 (1)
Peritonsillar abscess (Infections and infestations) | 0 | 1 (1) | 0
Pneumonia (Infections and infestations) | 1 (1) | 0 | 0
Tooth infection (Infections and infestations) | 1 (1) | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2) | 1 (1) | 0
Urosepsis (Infections and infestations) | 0 | 1 (2) | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 (1) | 2 (2)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 (1) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1 (1) | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 | 1 (1) | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 | 0
Liver function test increased (Investigations) | 0 | 1 (1) | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 10 (11) | 7 (7) | 3 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 3 (4)
Ketoacidosis (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 0
Ketosis (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0
Obesity (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 (1) | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 | 0
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 (1) | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 (1) | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 (1) | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 1 (1)
Cubital tunnel syndrome (Nervous system disorders) | 0 | 0 | 1 (1)
Hypoglycaemic seizure (Nervous system disorders) | 1 (1) | 0 | 0
Multiple sclerosis (Nervous system disorders) | 1 (1) | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 | 0
Adjustment disorder (Psychiatric disorders) | 0 | 0 | 1 (1)
Obstructive uropathy (Renal and urinary disorders) | 1 (1) | 0 | 0
Renal colic (Renal and urinary disorders) | 1 (1) | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 (1) | 0
Gynaecomastia (Reproductive system and breast disorders) | 1 (1) | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 1 (1) | 0
Embolism (Vascular disorders) | 0 | 0 | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 0 | 1 (1) | 0
Thrombosis (Vascular disorders) | 0 | 1 (2) | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin 5 mg + Insulin (N=277) | Dapagliflozin 10 mg + Insulin (N=296) | Placebo + Insulin (N=260)
Diarrhoea (Gastrointestinal disorders) | 11 (13) | 21 (25) | 9 (10)
Nausea (Gastrointestinal disorders) | 14 (18) | 15 (20) | 7 (7)
Gastroenteritis (Infections and infestations) | 15 (16) | 10 (13) | 8 (10)
Influenza (Infections and infestations) | 15 (18) | 15 (17) | 17 (23)
Upper respiratory tract infection (Infections and infestations) | 19 (26) | 28 (36) | 15 (28)
Urinary tract infection (Infections and infestations) | 27 (37) | 10 (12) | 19 (20)
Viral upper respiratory tract infection (Infections and infestations) | 51 (67) | 46 (65) | 48 (66)
Headache (Nervous system disorders) | 14 (17) | 20 (27) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an Investigator requests permission to publish data from this study any such publication is to be agreed with AstraZeneca (AZ) in advance. The investigator agrees to provide AZ as soon as possible with drafts of proposed publications. Unless otherwise agreed, AZ shall have a period of 60 days from receipt of the proposed final manuscript to review it and may within such time require that submission for publication of the manuscript be delayed in order for AZ to file patent applications.